CLINICAL TRIAL: NCT05593718
Title: Comparison of High-flow Nasal Oxygen Therapy and Face Mask Ventilation on Desaturations During Panendoscopy Under General Anesthesia
Brief Title: Comparison of HFNO and FMV on Desaturations During Panendoscopy Under General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, David Ferreira, Principal Investigator, Centre Hospitalier Universitaire de Besancon
Other Study IDs: ID052021HFNO
Record Dates: First submitted 2021-05-31; First posted 2022-10-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: ENT Tumor
Keywords: Panendoscopy; nasal high flow oxygen therapy; face mask ventilation; desaturation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FaceMask Ventilation (FMV): During the period from January 1, 2015, to December 31, 2016, all panendoscopies performed with FMV, whether urgent or scheduled and regardless of indication, were included. Panendoscopies performed with any other oxygenation method were excluded.
- HFNO: During the period from January 1, 2018, to December 31, 2019, all panendoscopies performed with HFNO, urgent or scheduled and regardless of indication, were included. Panendoscopies performed with any other oxygenation method were excluded.

SUMMARY:
Panendoscopy is a common procedure that requires deep and short anesthesia. The main challenge is the sharing of the airway between the anesthesia team and the surgical team. There are several methods to ensure oxygenation during this type of procedure: oro-tracheal intubation, jet ventilation, spontaneous ventilation anesthesia, apneic ventilation with intermittent face mask ventilation. There is no consensus regarding the best airway management technique for this procedure. Regardless of the method chosen to ensure oxygenation during this procedure, the risk of hypoxemia during desaturation episodes is significant.

However, the use of HFNO seems to show a prolongation of apnea time without desaturations (< 90% SpO2) and seems to allow the performance of panendocoscopies.

In the Besançon University Hospital, since 2017, all panendoscopies are performed with HFNO. Before 2017, panendoscopies were performed under face mask ventilation. The main of the study hypothesis is that HFNO brought a gain in terms of safety, especially on the desaturation rate compared to face mask ventilation.

The investigators will carry out a quasi-experimental study comparing two periods. The first period concerns the years 2015-2016. It aims to study patients who had panendoscopies performed under FMV. The second period covers the years 2018-2019. It aims to study patients who had panendoscopies performed under HFNO.

The year 2017 is considered as the washout period necessary to avoid the learning effect of the HFNO introduced during that year.

DETAILED DESCRIPTION:
Currently, there are several strategies to ensure oxygenation during this specific type of ENT management:

* Mechanical ventilation with oro-tracheal intubation (OTI)
* face mask ventilation (FMV)
* Jet ventilation
* HFNO Each of these methods has advantages and disadvantages, which explains why there are no clear recommendations to date on the preferred anesthesia and oxygenation technique. Regardless of the method chosen, the risks remain significant for the patient, particularly the risk of hypoxemia during a desaturation episode.

In 2017, HFNO was introduced for panendoscopies in the Besançon University Hospital. Before 2017, panendoscopies were mainly perfomed with intermittent face mask ventilation.

The objective of the study is to compare the FMV group (patients receiving panendoscopy and ventilated with FMV during 2015-2016) with the HFNO group (patients receiving panendoscopy and oxygenated with HFNO during 2018-2019) with respect to perprocedural hypoxemia (SpO2<90% for more than 1 minute).

Secondary objectives are to compare complications, use of oro-tracheal intubation, and procedure duration between the two oxygenation methods.

ELIGIBILITY:
Inclusion Criteria:

* major patients receiving panendoscopy
* patients ventilated by face mask during the first period,
* patients receiving oxygen by HFNO during the second period

Exclusion Criteria:

* Patients receiving ventilatory strategy other than those selected by time period.
* Patients receiving panendoscopies performed with a method of oxygenation other than those defined in their period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Face Mask Ventilation (FMV) Group :patients who had panendoscopies performed under FMV during the years 2015-2016.
  HFNO group :patients who had panendoscopies performed under HFNO during the years the years 2018-2019.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with oxygen desaturation | more than 1 minute during the intervention
  Proportion of patients with oxygen desaturation (SpO2 < 90%) for more than 1 minute.

SECONDARY OUTCOMES:
Proportion of patients requiring repeat face mask ventilation | more than 1 minute during the intervention
  Proportion of patients requiring repeat face mask ventilation (at least one reventilation outside the initial denitrogenation)
Proportion of patients requiring oro-tracheal intubation | during the intervention (max 6hours)from induction of anaesthesia to discharge from the operating theatre
  Proportion of patients intubated during panendoscopy
Duration of the procedure | during the intervention (max 6hours) from induction of anaesthesia to discharge from the operating theatre
  Time (minutes) from induction of anaesthesia to discharge from the operating theatre
Incidence of mild intraoperative complications | more than 1 minute during the intervention
  Complications are : mild bradycardia (between 45 and 30 beats per minute), hypotension defined by MAP (between 65 and 40mmHg), hypercapnia (betaween 60 and 80 mmHg)
Incidence of major intraoperative complications | more than 1 minute during the intervention
  Complications are : Tracheotomy, extreme bradycardia < 30 beats per minute, hemodynamic instability defined by MAP < 40mmHg, hypercapnia (more than 80 mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Besançon, Besançon, Franche Comté, France